CLINICAL TRIAL: NCT07003204
Title: Diagnostic and Prognostic Role of Pleural Fluid Neutrophil-to Lymphocyte and Monocyte-to-Lymphocyte Ratios in Exudative Pleural Effusion
Brief Title: Neutrophil-to Lymphocyte and Monocyte-to-Lymphocyte Ratios in Exudative Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Sabry, Lecturer of chest diseases, Alexandria University
Other Study IDs: lymphocyte- monocyte- exudate
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- only one group of patients: prospective cohort randomized control study
  Interventions: Procedure: medical thoracoscopy

INTERVENTIONS:
Procedure: medical thoracoscopy — pleural fluid aspiration and cellular analysis

SUMMARY:
Exudative pleural effusion (EPE) presents a diagnostic challenge, requiring accurate biomarkers to predict outcomes and guide treatment. The neutrophil-to-lymphocyte ratio (NLR) and monocyte-to-lymphocyte ratio (MLR) in pleural fluid are emerging as potential prognostic markers. We aimed to assess the diagnostic and prognostic utility of pleural fluid NLR and MLR in EPE.

DETAILED DESCRIPTION:
Pleural fluid NLR and MLR are reliable biomarkers for diagnosing malignant pleural effusion and predicting poorer survival outcomes. These ratios may be useful in clinical practice, especially in resource-limited settings, to guide decision-making in the management of pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18-80 years with an EPE diagnosis confirmed by thoracentesis.

Exclusion Criteria:

* Exclusion criteria included patients with a history of recent surgery, corticosteroid use, or those with mixed effusion types.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 person with pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-05-11 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
MLR and NLR measuring in pleural fluid | 1 month
  counting pleural fluid monocytes,lymphocytes and neutrophils

OTHER OUTCOMES:
MLR and NLR measuring in pleural fluid | one month
  counting the pleural monocytes, neutrophils and lymphoctes

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Sabry eltarhony, lecturer, Principal Investigator — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
not in the policy of the department

REFERENCES:
- See also: https://pmc.ncbi.nlm.nih.gov/articles/PMC8075197/ — https://pmc.ncbi.nlm.nih.gov/articles/PMC8075197/
- Available data/document: Clinical Study Report: msabry776@yahoo.com — https://pmc.ncbi.nlm.nih.gov/articles/PMC8075197/ — very good